CLINICAL TRIAL: NCT06077162
Title: Diabetes Nutrition Education (What Can I Eat? [WCIE]) and Healthy Food Resource for American Indians and Alaska Natives With T2D
Brief Title: Diabetes Nutrition Education and Healthy Food Resource for AIANs With T2D
Acronym: OKCICWCIE+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: American Diabetes Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other); Washington State University (Other); Oklahoma City Indian Clinic (Unknown); Gretchen Swanson Center for Nutrition (Other); University of North Carolina, Chapel Hill (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4595; 5K01DK128023 (NIH)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 3 arm RCT (nutrition education classes only, nutrition education classes + healthy food resource, healthy food resource only) - randomized at pt level, no stratification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- What Can I Eat Diabetes Nutrition Education Classes Only (Experimental): Participants will be enrolled in a 3 month, 5 session in-person diabetes nutrition education class, entitled What Can I Eat?, over the course of the 3 month intervention (4 * 90 min in person classes weekly for a month, with 5th class at 3 months from baseline).
  Interventions: Other: Diabetes Nutrition Education Classes
- What Can I Eat Diabetes Nutrition Education Classes + Healthy Food Security Resource (Experimental): Participants will be enrolled in a 3 month, 5 session in-person diabetes nutrition education class, entitled What Can I Eat?, over the course of the 3 month intervention (4 * 90 min in person classes weekly for a month, with 5th class at 3 months from baseline). Additionally, patients will receive a $30.00 healthy food resource weekly for 12 weeks.
  Interventions: Other: Diabetes Nutrition Education Classes; Other: Healthy Food Security Resource
- Healthy Food Security Resource Only (Experimental): Patients will receive a $30.00 healthy food resource weekly for 12 weeks.
  Interventions: Other: Healthy Food Security Resource

INTERVENTIONS:
Other: Diabetes Nutrition Education Classes — Diabetes nutrition education offered by registered dietitian in group-based classes.
  Arms: What Can I Eat Diabetes Nutrition Education Classes + Healthy Food Security Resource; What Can I Eat Diabetes Nutrition Education Classes Only
Other: Healthy Food Security Resource — Participants offered security resource which is a $30.00 Aldi (grocery store) gift card provided weekly for 12 weeks.
  Arms: Healthy Food Security Resource Only; What Can I Eat Diabetes Nutrition Education Classes + Healthy Food Security Resource

SUMMARY:
Healthy nutrition habits are key to managing type 2 diabetes (T2D). However, American Indian and Alaska Natives (AI/ANs) often lack access to culturally relevant nutrition education and they disproportionately experience food insecurity. Food insecurity, defined as lack of consistent access to enough food for an active, healthy life, negatively impacts one's ability to engage in diabetes self-management and care. The purpose of this study is to evaluate if diabetes nutrition education and an added food security resource, such as farmers market vouchers for fruits and vegetables, can improve diabetes self-management for AI/ANs with T2D. Researchers will work with collaborators at the Oklahoma City Indian Clinic in Oklahoma City, OK, and an American Indian community advisory board (CAB) throughout the study to ensure the nutrition education and food security resources are designed to meet the needs of the community and clinic. With the guidance of the CAB, researchers will recruit adults with T2D to participate in a 3-month intervention. Participants will be randomized into one of 3 groups. Some people will have diabetes nutrition education and the food security resource, some will have only the diabetes nutrition education, and some will receive only the food security resource. Outcomes such as food security status and clinical diabetes health indicators will be measured at 5 timepoints. This intervention is significant to diabetes because AI/ANs experience diabetes health disparities and the combination of diabetes nutrition education plus an added food security resource could help decrease T2D complications and improve quality of life for AI/ANs.

DETAILED DESCRIPTION:
Background: Healthy nutrition is key to T2D self-care and management. Culturally relevant nutrition education for American Indian and Alaska Natives (AI/Ans) is limited, contributing to diabetes health disparities, and disproportionate rates of food insecurity exacerbates these disparities.

Hypothesis: AI/ANs with T2D who receive both culturally relevant diabetes nutrition education and food security resources will have more improved outcomes (e.g., dietary intake, HbA1c) than AI/ANs with T2D who receive only diabetes nutrition education or a food security resource.

Supporting Rationale: Nutrition education improves T2D outcomes and reducing food insecurity can decrease diabetes health disparities.

Specific Aims: Aim #1: Engage an AI/AN community advisory board to support rigorous and equitable community based participatory research; Aim #2: Implement and evaluate a diabetes nutrition education and food security resource intervention in collaboration with the Oklahoma City Indian Clinic in Oklahoma City, OK.

Research Design: Three arm randomized controlled trial with: intervention group (diabetes nutrition education + food security resource); diabetes nutrition education group only; food security resource group only. Three month intervention with diabetes nutrition education and food security resource with 5 data collection timepoints: baseline, 1, 3, 6, 9 months. Outcomes include: HbA1c, blood pressure, dietary intake, diabetes distress, and food security.

Relevance to a cure, prevention and/or treatment of diabetes: Treatment of T2D among AI/ANs requires multi-level approaches to decrease health disparities related to social determinants of health such as lack of access to healthful foods. Providing both nutrition education and a food security resource could synergistically improve T2D self-management for AI/ANs

ELIGIBILITY:
Inclusion Criteria:

* Dx type 2 diabetes; American Indian or Alaska Native; fluent in English

Exclusion Criteria:

* Planned move within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 0, 3, 6, 9 months
  Participant HbA1c will be collected by point of care fingerstick or electronic medical record

SECONDARY OUTCOMES:
Blood pressure | 0, 3, 6, 9 months
  Participant systolic and diastolic blood pressure measurements collected by arm cuff automated BP read or electronic medical record
Body weight | 0, 3, 6, 9 months
  Body weight will be measured or collected via electronic medical record
Food insecurity | 0, 3, 6, 9 months
  Self reported survey: Food insecurity measured by 18 item USDA food security module
Diabetes distress | 0, 3, 6, 9 months
  Self reported survey: Participant diabetes distress measured by Problem Areas in Diabetes Scale (PAID-5)
Economic Quality of Life | 0, 3, 6, 9 months
  Self reported survey: 10 item measure assessing the economic quality of life
Perceived Diabetes Self Management Scale (PDSMS) | 0, 3, 6, 9 months
  Self reported survey: 8 item measure assessing perceived diabetes self management scale
What Can I Eat? Impact Survey | 0, 3, 6, 9 months
  Self reported survey: 30 item measure assessing knowledge, self efficacy, and behavior from participating in "What Can I Eat?" diabetes nutrition education
Dietary intake - 24 hour recall | 0, 3 months (2 * 24 hour recalls at each timepoint = 4 * 24 hour recalls per participant)
  Dietitian proctored 24 hour dietary recall using ASA24

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Stotz, PhD, Principal Investigator — Colorado State University
Locations (1):
- Oklahoma City Indian Clinic, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Tribes are sovereign Indian Nations that have a unique government-to-government relationship with the Federal government. Many discussions, publications, and treatises have addressed how this relationship affects the ownership and sharing of data. The growing consensus on the part of Tribal communities is that the Indian Nations have an inherent right to at least an equal say in the fate of raw data. More recently, these same rights have been exercised by community organizations and agencies serving Native peoples. Decisions about sharing of data cannot be made without full discussion and agreement by the participating tribes or agencies. Each Tribe involved must approve all provisions laid down in such policies prior to the release of data to any outside investigator or entity. This includes seeking approval for abstracts and manuscripts to be presented and submitted to academic or scientific conferences and journals.